CLINICAL TRIAL: NCT00135330
Title: An Evaluation of the Metabolic Effects of Exenatide, Rosiglitazone, and Exenatide Plus Rosiglitazone in Subjects With Type 2 Diabetes Mellitus Treated With Metformin
Brief Title: An Evaluation of Exenatide and Rosiglitazone in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-US-GWAY
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Results first posted 2009-08-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; exenatide; rosiglitazone; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide Arm (Experimental)
  Interventions: Drug: exenatide
- Exenatide plus Rosiglitazone Arm (Experimental)
  Interventions: Drug: exenatide; Drug: rosiglitazone
- Rosiglitazone Arm (Experimental)
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta
  Arms: Exenatide Arm; Exenatide plus Rosiglitazone Arm
Drug: rosiglitazone — oral tablet, 2mg or 4mg, twice a day
  Other Names: Avandia
  Arms: Exenatide plus Rosiglitazone Arm; Rosiglitazone Arm

SUMMARY:
This protocol is designed to evaluate the metabolic effects of adding exenatide, rosiglitazone, or both to an existing regimen of metformin in subjects with inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c of 6.8% to 10.0%, inclusive.
* Body mass index (BMI) of 25 kg/m^2 to 40 kg/m^2, inclusive.

Exclusion Criteria:

* Have participated in this study previously, or have received exenatide, pramlintide acetate, GLP-1 analogs, or dipeptidyl peptidase-IV (DPP-IV) inhibitors
* Have participated in an interventional, medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days of study start. This criterion includes drugs that have not received regulatory approval for any indication at the time of study start.
* Treated with any of the following medications:

  * Thiazolidinedione within 5 months of screening;
  * Sulfonylurea within 3 months of screening;
  * Metformin/sulfonylurea combination therapy within 3 months of screening;
  * Alpha-glucosidase inhibitor within 3 months of screening;
  * Meglitinide within 3 months of screening;
  * Insulin for more than 1 week within the 3 months prior to screening.
  * Symlin (pramlintide acetate) injection or Byetta (exenatide) injection at any time
  * Chronic (more than 2 weeks) or recent (within 4 weeks of study start) use of a drug that directly affects gastrointestinal motility
  * Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within the 4 weeks immediately preceding study start
  * Regular use of a medication with addictive potential such as an opiate, narcotic, or tranquilizer
  * Systemic antineoplastic agent
  * Systemic transplantation medication
  * Drugs for weight loss, including over-the-counter medications, within the 4 months prior to study start

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (19):
- United States (19):
  - Research Site, Phoenix, Arizona
  - Research Site, San Francisco, California
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, League City, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Renton, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] DeFronzo RA, Triplitt C, Qu Y, Lewis MS, Maggs D, Glass LC. Effects of exenatide plus rosiglitazone on beta-cell function and insulin sensitivity in subjects with type 2 diabetes on metformin. Diabetes Care. 2010 May;33(5):951-7. doi: 10.2337/dc09-1521. Epub 2010 Jan 27. PMID 20107105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between 18 October 2005 and 14 March 2008.
Groups:
- Exenatide: Exenatide 5 mcg twice a day (BID) for 4-weeks followed by exenatide 10 mcg BID for 16-weeks.
- Exenatide Plus Rosiglitazone: Exenatide 5 mcg BID + rosiglitazone 2 mg BID for 4-weeks followed by exenatide 10 mcg + rosiglitazone 4 mg BID for 16-weeks.
- Rosiglitazone: Rosiglitazone 2 mg BID for 4-weeks followed by rosiglitazone 4 mgs BID for 16-weeks.
Period: Overall Study
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Started | 45 | 47 | 45
Completed | 33 | 34 | 34
Not Completed | 12 | 13 | 11
Not completed — Adverse Event | 2 | 5 | 1
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Protocol Violation | 4 | 3 | 3
Not completed — Patient Decision | 5 | 1 | 4
Not completed — Sponsor Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone | Total
Number analyzed (Participants) | 45 | 47 | 45 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 37 | 36 | 109
  >=65 years | 9 | 10 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.99 (9.71) | 54.63 (9.91) | 55.54 (10.71) | 55.70 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 20 | 67
  Male | 23 | 22 | 25 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in ASIiAUC During a Hyperglycemic Clamp Test.
Description: Change in insulin incremental area under the concentration-time curve (ASIiAUC) from baseline to week 20. ASIiAUC is a measure of beta-cell function.
Time Frame: 20 weeks
Population: All patients in full analysis set who participated in clamp test and have both baseline and endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: uIU-min/ml
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 17 | 18 | 15
uIU-min/ml
  Baseline ASIiAUC | 643.40 (106.71) | 686.41 (103.70) | 786.12 (113.60)
  Change in ASIiAUC at week 20 | 747.26 (187.40) | 194.68 (181.59) | -99.85 (200.04)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; The ratio of the ASI-iAUC at Week 20 to that at baseline was compared between the treatment groups; Test type: Superiority or Other; p = 0.282, ANCOVA

2. Secondary Outcome: Change in AUC for Glucose During a Meal Challenge Test (MCT).
Description: Change in AUC(15-180 min) for glucose during a MCT baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who have both baseline and endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: mmol-min/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 35 | 34
mmol-min/L
  Baseline glucose AUC during MCT | 1782.86 (60.47) | 1799.68 (59.60) | 1741.87 (60.47)
  Change in glucose AUC during MCT at week 20 | -560.12 (50.95) | -635.24 (50.25) | -425.59 (51.02)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.004, ANCOVA

3. Secondary Outcome: Change in Insulin Sensitivity Index as Measured by M-value.
Description: Change of M-Value (mg/kg-min) during hyperinsulinemic euglycemic clamp test from baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who participated in clamp test and have both baseline and endpoint measurements.
Measure: Least Squares Mean (Standard Error); unit: mg/kg-min
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 16 | 16 | 15
mg/kg-min
  M-Value at baseline | 3.89 (0.495) | 2.49 (0.495) | 4.02 (0.511)
  Change in M-Value from baseline at week 20 | 0.477 (0.425) | 2.07 (0.440) | 1.42 (0.442)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.308, ANCOVA

4. Secondary Outcome: Change in Insulin AUC in the First Stage From Baseline to Endpoint.
Description: Change in insulin AUC in the first stage(uIU-min/ml) from baseline to week 20. "First stage" represents the first 10 minutes after reaching a steady state during a hyperglycemic clamp test.
Time Frame: Week 20
Population: All patients in full analysis set who participated in clamp tests and have both baseline and endpoint
Measure: Least Squares Mean (Standard Error); unit: uIU-min/ml
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 17 | 17 | 15
uIU-min/ml
  Baseline insulin AUC | 200.50 (50.40) | 136.84 (50.40) | 157.49 (53.66)
  Change from baseline insulin AUC at week 20 | 134.88 (31.71) | 32.12 (31.65) | -50.81 (33.59)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.079, ANCOVA

5. Secondary Outcome: Change in Insulin iAUC From Baseline to Endpoint.
Description: Change in insulin iAUC in the first stage(uIU-min/ml) from baseline to week 20. "First stage" represents the first 10 minutes after reaching a steady state during a hyperglycemic clamp test.
Time Frame: Week 20
Population: All patients in full analysis set who participated in clamp tests and have both baseline and endpoint.
Measure: Least Squares Mean (Standard Error); unit: uIU-min/ml
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 17 | 17 | 15
uIU-min/ml
  Baseline insulin iAUC | 5.98 (14.29) | -9.92 (14.29) | 23.09 (15.21)
  Change from baseline insulin iAUC at week 20 | 99.08 (24.23) | 53.71 (24.54) | 11.51 (26.15)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.252, ANCOVA

6. Secondary Outcome: Ratio (Value at Endpoint Divided by Value at Baseline) of AUC for Insulin During a Meal Challenge Test (MCT).
Description: Ratio (value at endpoint divided by value at baseline) of AUC (15-180 min) for insulin (uIU-min/ml) during MCT.
Time Frame: Week 20
Population: All patients in full analysis set who have both baseline and endpoint measurement.
Measure: Geometric Mean (Standard Error); unit: uIU-min/ml
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 35 | 33
uIU-min/ml
  Baseline AUC for insulin during MCT | 5171.40 (522.82) | 4324.13 (430.87) | 5816.83 (596.91)
  Ratio(endpoint/baseline) of insulin AUC during MCT | 0.806 (0.063) | 0.664 (0.052) | 0.722 (0.058)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.465, ANCOVA

7. Secondary Outcome: Change in AUC for C-peptide During a Meal Challenge Test (MCT).
Description: Ratio (value at endpoint divided by value at baseline) of AUC(15-180 min) for C-peptide (nmol-min/L) during a MCT from baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who have both baseline and endpoint measurement.
Measure: Geometric Mean (Standard Error); unit: nmol-min/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 34 | 32
nmol-min/L
  Baseline C-peptide during a MCT | 319.77 (18.13) | 310.51 (17.61) | 325.65 (19.04)
  Ratio(endpoint/baseline) of C-peptide during a MCT | 0.908 (0.040) | 0.804 (0.036) | 0.854 (0.039)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.348, ANCOVA

8. Secondary Outcome: Change in Incremental for Postprandial Glucose During a Meal Challenge Test (MCT).
Description: Change in incremental for postprandial glucose (mmol/L) during a MCT from baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who have both baseline and endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 34 | 33
mmol/L
  Baseline glucose at 15 min | 0.950 (0.138) | 1.12 (0.138) | 0.828 (0.142)
  Change fr baseline glucose at 15 min at wk 20 | -0.651 (0.151) | -0.286 (0.152) | 0.150 (0.157)
  Baseline glucose at 30 min | 2.39 (0.218) | 2.54 (0.221) | 2.23 (0.221)
  Change fr baseline glucose at 30 min at wk 20 | -1.46 (0.248) | -1.06 (0.252) | -0.066 (0.252)
  Baseline glucose at 60 minutes | 3.59 (0.273) | 3.88 (0.273) | 3.48 (0.273)
  Change fr baseline glucose at 60 min at wk 20 | -2.56 (0.329) | -2.46 (0.330) | -0.720 (0.329)
  Baseline glucose at 90 minutes | 3.24 (0.231) | 3.36 (0.228) | 3.48 (0.239)
  Change fr baseline glucose at 90 min at wk 20 | -2.87 (0.312) | -2.91 (0.307) | -0.952 (0.322)
  Baseline glucose at 120 minutes | 2.49 (0.235) | 2.24 (0.238) | 2.31 (0.235)
  Change fr baseline glucose at 120 min at wk 20 | -2.24 (0.271) | -2.52 (0.275) | -0.912 (0.271)
  Baseline glucose at 150 minutes | 1.62 (0.230) | 1.14 (0.230) | 1.25 (0.230)
  Change fr baseline glucose at 150 min at wk 20 | -1.42 (0.288) | -1.95 (0.287) | -0.830 (0.286)
  Baseline glucose at 180 minutes | 0.461 (0.235) | 0.036 (0.235) | 0.279 (0.235)
  Change fr baseline glucose at 180 min at wk 20 | -0.583 (0.231) | -0.995 (0.232) | -0.481 (0.230)

9. Secondary Outcome: Change in Incremental for Postprandial Insulin During Meal Challenge Test (MCT).
Description: Change in incremental for postprandial insulin (mmol/L) during meal challenge test (MCT) from baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who have both baseline and endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 35 | 32
mmol/L
  Baseline insulin at 15 min | 9.97 (1.71) | 8.09 (1.71) | 7.53 (1.79)
  Change fr baseline insulin at 15 min at wk 20 | -1.71 (1.45) | -1.84 (1.45) | -0.455 (1.52)
  Baseline insulin at 30 min | 19.81 (2.28) | 14.79 (2.25) | 18.83 (2.35)
  Change fr baseline insulin at 30 min at wk 20 | -3.00 (1.90) | -2.63 (1.89) | -1.04 (1.96)
  Baseline insulin at 60 min | 27.92 (4.68) | 27.67 (4.61) | 32.09 (4.75)
  Change fr baseline insulin at 60 min at wk 20 | -11.04 (2.63) | -7.47 (2.59) | -7.42 (2.67)
  Baseline insulin at 90 min | 26.06 (4.10) | 21.85 (4.10) | 32.25 (4.36)
  Change fr baseline insulin at 90 min at wk 20 | -9.42 (2.72) | -9.27 (2.74) | -6.19 (2.92)
  Baseline insulin at 120 min | 19.56 (2.99) | 17.52 (2.99) | 25.47 (3.04)
  Change fr baseline insulin at 120 min at wk 20 | -11.26 (1.99) | -8.69 (2.00) | -6.43 (2.04)
  Baseline insulin at 150 min | 15.67 (2.47) | 12.74 (2.43) | 18.11 (2.51)
  Change fr baseline insulin at 150 min at wk 20 | -7.48 (1.74) | -8.13 (1.73) | -5.57 (1.78)
  Baseline insulin at 180 min | 10.58 (1.73) | 8.18 (1.73) | 10.74 (1.79)
  Change fr baseline insulin at 180 min at wk 20 | 0.031 (1.30) | -5.26 (1.30) | -4.04 (1.34)

10. Secondary Outcome: Change in Incremental for Postprandial C-peptide During Meal Challenge Test (MCT).
Description: Change in incremental for postprandial C-peptide (mmol/L) during MCT from baseline to week 20.
Time Frame: Week 20
Population: All patients in full analysis set who have baseline and endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 34 | 32
mmol/L
  Baseline C-peptide at 15 min | 0.238 (0.049) | 0.259 (0.049) | 0.206 (0.051)
  Change fr baseline C-peptide at 15 min at week 20 | -0.006 (0.045) | 0.016 (0.046) | 0.087 (0.047)
  Baseline C-peptide at 30 min | 0.521 (0.059) | 0.517 (0.059) | 0.560 (0.061)
  Change fr baseline C-peptide at 30 min at week 20 | -0.071 (0.056) | -0.036 (0.056) | 0.099 (0.058)
  Baseline C-peptide at 60 min | 0.818 (0.110) | 0.871 (0.110) | 0.881 (0.114)
  Change fr baseline C-peptide at 60 min at week 20 | -0.148 (0.090) | -0.025 (0.090) | 0.054 (0.093)
  Baseline C-peptide at 90 min | 0.895 (0.100) | 0.953 (0.101) | 1.03 (0.106)
  Change fr baseline C-peptide at 90 min at week 20 | -0.185 (0.099) | -0.117 (0.101) | -0.052 (0.106)
  Baseline C-peptide at 120 min | 0.817 (0.112) | 0.828 (0.114) | 0.972 (0.114)
  Change fr baseline C-peptide at 120 min at week 20 | -0.259 (0.100) | -0.134 (0.102) | -0.016 (0.102)
  Baseline C-peptide at 150 min | 0.843 (0.091) | 0.651 (0.091) | 0.813 (0.092)
  Change fr baseline C-peptide at 150 min at week 20 | -0.251 (0.095) | -0.254 (0.095) | -0.093 (0.096)
  Baseline C-peptide at 180 min | 0.610 (0.084) | 0.482 (0.085) | 0.619 (0.087)
  Change fr baseline C-peptide at 180 min at week 20 | -0.075 (0.062) | -0.238 (0.063) | -0.092 (0.064)

11. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 35 | 36 | 34
Percentage
  Baseline HbA1c | 7.79 (0.116) | 7.84 (0.115) | 7.92 (0.116)
  Change from baseline HbA1c at week 20 | -0.908 (0.118) | -1.31 (0.116) | -0.968 (0.118)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.039, Mixed Model Repeated Measures (MMRM)

12. Secondary Outcome: Change in Fasting Serum Glucose Concentration.
Description: Change in fasting serum glucose concentration from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 35 | 34
mmol/L
  Baseline fasting serum glucose | 8.42 (0.278) | 8.43 (0.271) | 8.48 (0.274)
  Change fr baseline fasting serum glucose at wk 20 | -1.46 (0.250) | -1.60 (0.244) | -1.80 (0.250)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.555, MMRM

13. Secondary Outcome: Change in Fasting C-peptide
Description: Change in fasting C-peptide from baseline to week 20.
Time Frame: Week 20
Population: Fasting C-peptide was initially identified as an outcome measure, but data for this measure were not subsequently collected at baseline or endpoint.
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change in Fasting Insulin
Description: Change in fasting insulin from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Geometric Mean (Standard Error); unit: uIU/ml
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 35 | 35 | 31
uIU/ml
  Baseline fasting insulin | 12.84 (1.55) | 10.96 (1.33) | 12.77 (1.54)
  Ratio (wk20/baseline)of fasting insulin | 0.980 (0.096) | 0.599 (0.059) | 0.755 (0.078)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.106, MMRM

15. Secondary Outcome: Change in Fasting Proinsulin
Description: Ratio (endpoint value divided by baseline value) for fasting proinsulin, comparing endpoint (week 20) to baseline
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Geometric Mean (Standard Error); unit: pmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 34 | 33
pmol/L
  Baseline fasting proinsulin | 4.32 (0.523) | 3.80 (0.455) | 3.56 (0.423)
  Ratio(wk20/baseline)of fasting proinsulin | 0.663 (0.073) | 0.538 (0.058) | 0.623 (0.068)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.341, MMRM

16. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 20.
Time Frame: Week 20
Population: All patients who aave both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 44 | 45 | 44
kg
  Baseline body weight | 93.05 (2.39) | 93.76 (2.36) | 91.78 (2.39)
  Change in body weight at week 20 | -2.82 (0.547) | -1.21 (0.538) | 1.48 (0.547)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p < 0.001, MMRM

17. Secondary Outcome: Change in Fasting Total Cholesterol.
Description: Change in fasting total cholestrol from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 36 | 34
mmol/L
  Baseline total cholesterol | 4.42 (0.150) | 4.41 (0.145) | 4.62 (0.149)
  Change fr baseline total cholesterol at week 20 | -0.128 (0.118) | 0.258 (0.114) | 0.438 (0.118)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.276, MMRM

18. Secondary Outcome: Change in Fasting HDL Cholesterol
Description: Change in fasting high-density lipoprotein (HDL) cholesterol from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 36 | 34
mmol/L
  Baseline HDL | 1.13 (0.048) | 1.17 (0.047) | 1.17 (0.048)
  Change from baseline HDL at week 20 | 0.022 (0.030) | 0.046 (0.029) | 0.055 (0.030)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.840, MMRM

19. Secondary Outcome: Change in Fasting LDL Cholesterol
Description: Change in fasting low-density lipoprotein (LDL) cholesterol from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 35 | 34
mmol/L
  Baseline LDL | 2.59 (0.131) | 2.57 (0.128) | 2.71 (0.129)
  Change from baseline LDL at week 20 | -0.049 (0.102) | 0.096 (0.100) | 0.334 (0.101)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.096, MMRM

20. Secondary Outcome: Change in Fasting Triglycerides
Description: Ratio (endpint value divided by baseline value) of fasting triglycerides from baseline to week 20.
Time Frame: Week 20
Population: All patients who have both baseline and at least one post baseline value in full analysis set
Measure: Geometric Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 34 | 36 | 34
mmol/L
  Baseline triglyceride | 1.56 (0.124) | 1.67 (0.128) | 1.76 (0.138)
  Ratio (endpoint/baseline) for triglycerides | 0.861 (0.060) | 0.977 (0.066) | 0.992 (0.069)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.875, MMRM

21. Secondary Outcome: Change in Percent Body Fat During a Meal Challenge Test (MCT)
Description: Change in percent body fat from baseline to week 20, as assessed during an MCT
Time Frame: 20 weeks
Population: All Patients in Full Analysis Set Who Have Both Baseline and Endpoint Measurement
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 34 | 32
percentage
  Baseline percent body fat | 33.42 (1.16) | 34.07 (1.15) | 32.50 (1.18)
  Change in percent body fat at week 20 | -1.40 (1.06) | -0.347 (1.04) | -1.18 (1.08)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.581, ANCOVA

22. Secondary Outcome: Change in Body Fat Mass During a Meal Challenge Test (MCT)
Description: Change in body fat mass form baseline to week 20, as assessed during an MCT
Time Frame: 20 weeks
Population: All Patients in Full Analysis Set Who Have Both Baseline and Endpoint Measurements
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 34 | 32
kg
  Baseline body fat mass | 32.05 (1.64) | 32.55 (1.62) | 30.54 (1.67)
  Change in body fat mass at week 20 | -2.76 (1.37) | -1.06 (1.35) | -1.99 (1.40)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.631, ANCOVA

23. Secondary Outcome: Change in Lean Body Mass During a Meal Challenge Test (MCT)
Description: Change in lean body mass from baseline to week 20, as assessed during an MCT
Time Frame: 20 weeks
Population: All Patients in Full Analysis Set Who Have Both Baseline and Endpoint Measurements
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 34 | 32
kg
  Baseline lean body mass | 64.62 (2.11) | 60.94 (2.08) | 61.09 (2.14)
  Change in lean body mass at week 20 | -2.99 (1.39) | 0.532 (1.37) | 1.23 (1.41)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.724, ANCOVA

24. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline to week 20
Time Frame: 20 weeks
Population: All Patients Who Have Both Baseline and At Least One Post Baseline Value in Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 35 | 33
cm
  Baseline waist circumference | 105.98 (1.68) | 106.85 (1.67) | 105.34 (1.67)
  Change in waist circumference at Week 20 | -2.95 (0.975) | -2.38 (0.955) | -0.225 (0.969)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.117, MMRM

25. Secondary Outcome: Change in Hip Circumference
Description: Change in hip circumference form baseline to week 20
Time Frame: 20 weeks
Population: All Patients Who Have Both Baseline and At Least One Post Baseline Value in Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 35 | 33
cm
  Baseline hip circumference | 113.29 (1.71) | 112.12 (1.69) | 111.90 (1.69)
  Change in hip circumference at week 20 | -1.28 (0.848) | 0.147 (0.827) | 1.51 (0.838)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.251, MMRM

26. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Change in waist-to-hip ratio (waist circumference divided by hip circumference) from baseline to week 20
Time Frame: 20 weeks
Population: All Patients Who Have Both Baseline and At Least One Post Baseline Value in Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: ratio (cm/cm)
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 33 | 35 | 33
ratio (cm/cm)
  Baseline waist-to-hip ratio | 0.939 (0.012) | 0.957 (0.012) | 0.943 (0.012)
  Change in waist-to-hip ratio at week 20 | -0.016 (0.011) | -0.022 (0.010) | -0.016 (0.011)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.710, MMRM

27. Secondary Outcome: Incidence of Hypoglycemia Events
Description: Number of subjects experiencing hypoglycemia at any point during the study
Time Frame: 20 weeks
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 45 | 47 | 45
participants | 8 | 9 | 6
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.575, Fisher Exact

28. Secondary Outcome: Hypoglycemia Rate Per 30 Days Per Patient
Description: Average number of episodes of hypoglycemia per 30 days per patient
Time Frame: 20 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hypoglycemia events / 30 days / patient
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 45 | 47 | 45
hypoglycemia events / 30 days / patient | 0.391 (0.298) | 0.594 (0.436) | 0.853 (1.05)
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.436, ANOVA

29. Secondary Outcome: Pedal Edema Score
Description: Pedal edema scores experienced by each patient throughout the study ("1+" indicates a patient experienced a pedal edema score of 1 , 2, or 3; "2+" indicates a patient experienced a pedal edema score of 2 or 3, etc.)
  Scale:
  1. Slight pitting, no visible distortion, disappears rapidly
  2. A somewhat deeper pit than in 1+, but again no readily detectable distortion, and it disappears in 10 - 15 seconds
  3. The pit is noticeably deep and may last more than a minute; the dependent extremity looks fuller and swollen
  4. The pit is very deep, lasts as long as 2 - 5 minutes, and the dependent extremity is grossly distorted
Time Frame: 20 weeks
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Number analyzed (Participants) | 44 | 45 | 44
participants
  No edema | 37 | 34 | 30
  Edema score: 1+ | 7 | 11 | 14
  Edema score: 2+ | 1 | 3 | 6
  Edema score: 3+ | 0 | 0 | 1
Statistical Analysis 1: Comparison: Exenatide Plus Rosiglitazone vs Rosiglitazone; Test type: Superiority or Other; p = 0.168, Generalized Linear Model

ADVERSE EVENTS:
Arm/Group | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Serious Adverse Events (participants affected / at risk) | 3 | 4 | 4
Other Adverse Events (participants affected / at risk) | 35 | 41 | 33
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/45 | 1/47 | 0/45
Cellulitis (Infections and infestations) | 0/45 | 0/47 | 1/45
Chest pain (Musculoskeletal and connective tissue disorders) | 1/45 | 0/47 | 0/45
Colitis ischaemic (Gastrointestinal disorders) | 0/45 | 1/47 | 0/45
Diverticulitis (Infections and infestations) | 0/45 | 0/47 | 1/45
Gastroenteritis (Infections and infestations) | 1/45 | 0/47 | 0/45
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/45 | 0/47 | 1/45
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/45 | 0/47 | 0/45
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1/45 | 0/47 | 0/45
Helicobacter gastritis (Infections and infestations) | 1/45 | 0/47 | 0/45
Major depression (Psychiatric disorders) | 0/45 | 1/47 | 0/45
Osteomyelitis (Infections and infestations) | 0/45 | 0/47 | 1/45
Otitis externa (Infections and infestations) | 0/45 | 1/47 | 0/45
Renal failure acute (Renal and urinary disorders) | 0/45 | 0/47 | 1/45
Staphylococcal infection (Infections and infestations) | 1/45 | 0/47 | 0/45
Suicidal ideation (Psychiatric disorders) | 0/45 | 1/47 | 0/45
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/45 | 0/47 | 1/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide | Exenatide Plus Rosiglitazone | Rosiglitazone
Nausea (Gastrointestinal disorders) | 21/45 | 22/47 | 2/45
Vomiting (Gastrointestinal disorders) | 10/45 | 9/47 | 0/45
Dizziness (Nervous system disorders) | 6/45 | 7/47 | 3/45
Oedema peripheral (General disorders) | 2/45 | 5/47 | 9/45
Diarrhoea (Gastrointestinal disorders) | 3/45 | 10/47 | 2/45
Headache (Nervous system disorders) | 5/45 | 4/47 | 3/45
Contusion (Injury, poisoning and procedural complications) | 3/45 | 5/47 | 2/45
Fatigue (General disorders) | 5/45 | 1/47 | 2/45
Upper respiratory tract infection (Infections and infestations) | 3/45 | 1/47 | 4/45
Injection site bruising (General disorders) | 3/45 | 4/47 | 0/45
Asthenia (General disorders) | 2/45 | 3/47 | 1/45
Anaemia (Blood and lymphatic system disorders) | 1/45 | 1/47 | 3/45
Constipation (Gastrointestinal disorders) | 2/45 | 3/47 | 0/45
Flatulence (Gastrointestinal disorders) | 2/45 | 3/47 | 0/45
Hunger (General disorders) | 3/45 | 1/47 | 0/45
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3/45 | 1/47 | 0/45
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/45 | 0/47 | 3/45
Diverticulitis (Infections and infestations) | 0/45 | 0/47 | 3/45
Oedema (General disorders) | 0/45 | 0/47 | 3/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days